CLINICAL TRIAL: NCT02865317
Title: Investigating the Long-Term Cortical Effects of Peripheral Nerve Injury At Birth
Brief Title: Cortical Effects of Peripheral Nerve Injury At Birth
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Gazi University (Other)
Collaborators: Ataturk Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Zeynep Tuna, Principal Investigator, Gazi University
Other Study IDs: GaziU-ZTuna1
Record Dates: First submitted 2016-01-29; First posted 2016-08-12 (Estimated); Last update posted 2016-08-12 (Estimated); Status verified 2016-08

CONDITIONS: Peripheral Nerve Injury
MeSH Terms: conditions — Peripheral Nerve Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Study group: Patients with obstetrical brachial plexus injury involving upper trunk (C5-6)

SUMMARY:
Cortical activity during rest and with stimulation by functional magnetic resonance imaging will be investigated in patients with OBPI.

DETAILED DESCRIPTION:
Peripheral nerve injury results in a number of cortical changes due to the lack of sensory and motor stimuli. Although functional magnetic resonance imaging (fMRI) studies that revealed the changes in the cortical activation exist, the cortical activation changes in obstetrical brachial plexus injury is poorly known. For this reason, the aim of this study is to investigate the cortical activity during rest and with stimulation by fMRI in patients with OBPI.

Patients with OBPI diagnosis in the cervical 5-6 (C5-6) (upper trunk) who are followed up in Gazi University Faculty of Health Sciences Department of Physiotherapy and Rehabilitation Division of Hand Rehabilitation will participate in the study. Patients with a surgery history at least 5 years ago and over 10 years age will be included. Clinical motor and sensory assessments will be performed to help in explaining the analyses of cortical activation. In their first visit, clinical assessments including Active Movement Scale, modified Mallet Classification (MMC) and sensory tests will be performed; while fMRI scanning will be carried out in the second visit. Patients will be scanned for 3 paradigms at one single fMRI session: at rest and during sensory stimulation and watching videos of motor movements. Video images will include the 5 movements used in MMC and will be watched by glasses integrated in the MRI device. Images obtained from MR scanning will be analyzed with analysis programs like Leonardo, Fresurfer, SPM, BrainVoyager and clinical results will be compared to MR images.

ELIGIBILITY:
Inclusion Criteria:

* upper trunk (cervical 5-6) involvement
* cooperated

Exclusion Criteria:

* illiterate
* surgical history for his arm in the previous 5 years
* other than only C5-6 involvement
* any impairment that prevents positioning in MRI machine

Ages: 10 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with obstetrical brachial plexus palsy
Sampling Method: Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2016-10; Primary Completion 2016-12 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
voxels | 6 months
  voxels (n) are the task-activated volume of brain regions

SECONDARY OUTCOMES:
Active Movement Scale score | 6 months
  AMS is a clinical outcome measure that evaluates patient's affected arm movements.This tool is used to quantify upper extremity strength by observing spontaneous, active movement both without and against gravity.

IPD SHARING:
Plan to Share IPD: No